CLINICAL TRIAL: NCT03032237
Title: Testing the Effectiveness and Acceptance of Home-delivered Protein-rich Meals and Foods on the Intake of Community-dwelling Older Adults.
Brief Title: Increase Protein Intake of Older Meal Service Clients With Readymade Protein-rich Meals and Foods
Acronym: ConsuMEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN University of Applied Sciences (Other)
Collaborators: HAS Hogeschool (Unknown); Centre of Expertise Food (CoE Food) (Unknown); Sligro (Unknown); FrieslandCampina (Industry)
Responsible Party: Principal Investigator, dr. Marian de van der Schueren, Prof. Dr., HAN University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ConsuMEER onderzoek
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Malnutrition; Protein; Protein Malnutrition
Keywords: Protein intake; Older adults; Protein-rich; Acceptance; Liking; Readymade meals
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-rich assortment (Experimental): The intervention groups receives protein-rich meals and protein-rich dairy products.
  Interventions: Other: Nutritional intervention - protein-rich
- Standard assortment (Placebo Comparator): The control group receives standard meals and food products.
  Interventions: Other: Nutritional intervention - standard

INTERVENTIONS:
Other: Nutritional intervention - protein-rich — Both groups will receive readymade meals (Sligro) for each day during the 4-week intervention period (28 hot meals in total per participant). They will also receive other food products from FrieslandCampina's assortment to freely consume during the intervention period.
  To keep the intervention as close as possible to the real life situation, meals and foods will be home-delivered twice a week as the participants are already used to.
  Intervention group will receive protein-rich meals and protein-rich foods and drinks.
  Arms: Protein-rich assortment
Other: Nutritional intervention - standard — Both groups will receive readymade meals (Sligro) for each day during the 4-week intervention period (28 hot meals in total per participant). They will also receive other food products from FrieslandCampina's assortment to freely consume during the intervention period.
  To keep the intervention as close as possible to the real life situation, meals and foods will be home-delivered twice a week as the participants are already used to.
  Control group will receive standard (not protein-rich) meals and standard foods and drinks.
  Arms: Standard assortment

SUMMARY:
Rationale: Undernutrition risk among community-dwelling older adults in developed countries is shown to be around 24%. Increasing protein intake is a strategy that is feasible as well as efficacious to reduce undernutrition in community-dwelling older adults. A promising strategy to increase protein intake among older adults, is to offer dietary solutions with normal foods that fit their current daily eating patterns. For this reason, home-delivered protein-rich readymade meals and protein-rich dairy products will be studied in this research.

Objective: The primary objective is to study the effectiveness of commercially available protein-rich readymade meals and protein-rich dairy products in increasing protein intake of older adults who use a meal-delivery service to a level of 1.2 g/kg bodyweight/d. Secondary objectives include: studying effects of these meals and dairy products on total daily energy intake. Further, studying the acceptance of and compliance to the meals and dairy products.

Study design: The study will be performed as a single-blind randomized, controlled, four-week trial in a real-life setting: in community-dwelling older adults' own homes.

Study population: The target group of this study are community-dwelling older adults who use a meal-delivery service.

Intervention: Both groups will receive readymade meals for each day during 4 weeks. They will also receive dairy products to freely consume during the intervention period. The intervention groups receives protein-rich meals and protein-rich dairy products, the control receives standard meals and food products.

Main study parameters/endpoints: Difference in daily protein intake between intervention and control group. Secondary parameters: energy intake and acceptance (liking).

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or over
* Living at home
* Be a client of maaltijdservice.nl
* Being able to eat by themselves
* Have a microwave to heat meals
* Live in Nijmegen or Den Bosch area
* Being able to understand, read and speak Dutch
* Having signed informed consent.

Exclusion Criteria:

* Legally incapacitated
* Mini Mental State Examination (MMSE) score < 24
* Following a diet with protein restriction or a vegetarian diet
* Allergies or intolerances prohibiting the use of dairy products
* Only using texture modified foods (liquid diet)
* Diagnosed by doctor with renal insufficiency
* Suffering from a terminal illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Protein intake | 4 weeks
  Difference in daily protein intake between intervention and control group assessed with 3-day food records which will be checked by trained dietitians.

SECONDARY OUTCOMES:
Acceptance | 4 weeks
  Acceptance and liking of meals and food products; outcome will be measured with a questionnaire including a 5-point likert scale (for liking) and a question how much was eaten. This questionnaire needs to be done every day.
Energy intake | 4 weeks
  Difference in daily energy intake between intervention and control group assessed with 3-day food records which will be checked by trained dietitians.

CONTACTS AND LOCATIONS:
Overall Officials: Marian de van der Schueren, PhD, Principal Investigator — HAN University of Applied Sciences; Annet Roodenburg, PhD, Principal Investigator — HAS Hogeschool
Locations (1):
- HAN University of Applied Sciences, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.